CLINICAL TRIAL: NCT05796479
Title: A 2-part, Open Label, Phase 1 Study to Investigate the Pharmacokinetics, Safety and Tolerability of Two Different Amlitelimab Drug Products After Administration of a Single Subcutaneous Dose in Healthy Adult Participants
Brief Title: A PK Comparability Study of Two Different Amlitelimab Drug Products in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PKM17597
Record Dates: First submitted 2023-03-13; First posted 2023-04-03 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: 2-part, open-label study with 1 arm in Part 1 and a randomized, 2 arms parallel design in Part 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Part1) (Experimental): Participants will receive a single SC dose of amlitelimab DP1 on Day 1.
  Interventions: Drug: Amlitelimab DP1
- Group 2 (Part 2) (Experimental): Participants will receive a single SC dose of amlitelimab DP1 on Day 1.
  Interventions: Drug: Amlitelimab DP1
- Group 3 (Part 2) (Experimental): Participants will receive a single SC dose of amlitelimab DP2 on Day 1.
  Interventions: Drug: Amlitelimab DP2

INTERVENTIONS:
Drug: Amlitelimab DP1 — Injection solution 1
  Subcutaneous
  Arms: Group 1 (Part1); Group 2 (Part 2)
Drug: Amlitelimab DP2 — Injection solution 2
  Subcutaneous
  Arms: Group 3 (Part 2)

SUMMARY:
This is a 2-part, Phase 1 study, with 1 arm in Part 1 and a randomized parallel design in Part 2. The purpose of this study is to evaluate the comparability of pharmacokinetics, safety and tolerability of two different amlitelimab drug products (DPs) after administration of a single subcutaneus (SC) dose in healthy adult participants.

Study details include:

The study duration for a participant will be approximately 17 weeks. The study includes a screening period of up to 28 days, a 4-day institutionalization period, and a follow up period for approximately 89 days (9 visits).

DETAILED DESCRIPTION:
The study duration for a participant will be approximately 17 weeks

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, ECG, and laboratory tests
* Body weight within 55 to 100 kg and body mass index (BMI) within the range 18-30 kg/m2 (inclusive)
* Male or female of childbearing potential are required to either practice true abstinence consistent with their preferred and usual lifestyle or use highly effective contraceptive methods for the entire duration of the treatment until 4 months after the investigational medicinal product (IMP) dosing.

Exclusion Criteria:

* Any history or presence of clinically relevant immunologic, cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness, unless the investigator considers an abnormality to be not clinically significant.
* Participants with a history of helminthic infection or invasive opportunistic infections such as histoplasmosis, listeriosis, coccidioidomycosis, candidiasis, Pneumocystis jirovecii, aspergillosis, irrespective of resolution.
* Serious infections requiring hospitalization within 30 days prior to screening or any active infection requiring treatment during screening.
* Current or past diagnosis of malignancies within the last 5 years prior to screening (except documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ).
* Presence or history of drug hypersensitivity or allergic disease diagnosed and treated by a physician.
* Evidence of active or latent tuberculosis (TB XE ' TB ' \f Abbreviation \t 'tuberculosis ' ) as documented by medical history and examination; TB testing via a positive (not indeterminate) QuantiFERON TB Gold test
* If female, pregnancy (defined as positive beta human chorionic gonadotropin [β-HCG] test), or lactating. - Received a live (attenuated) immunization within 12 weeks prior to inclusion or non-live immunization within 4 weeks prior to inclusion.
* Any medication, with the exception of hormonal contraception, within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, whichever is longer, and any biologics (antibody or its derivatives) given within 4 months before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Plasma concentration observed (Cmax ) | From Day1 up to Day92 (end of study [EOS])
  Cmax after administration of a single SC dose of amlitelimab DP 1
Part 1: Area under the curve from the time of dosing to the last measurable concentration (AUClast) | From Day1 up to Day92 (EOS)
  AUClast after administration of a single SC dose of amlitelimab DP 1
Part 1: Area under the plasma concentration versus time curve extrapolated to infinity (AUC) | From Day1 up to Day92 (EOS)
  AUC after administration of a single SC dose of amlitelimab DP 1
Part 2: Cmax of two different amlitelimab DPs (DP1 and DP2) | From Day1 up to Day92 (EOS)
  Cmax after administration of a single SC dose of amlitelimab DP 1 and DP2
Part 2: AUClast of two different amlitelimab DPs (DP1 and DP2) | From Day1 up to Day92 (EOS)
  AUClast after administration of a single SC dose of amlitelimab DP1 and DP 2
Part 2: AUC of two different amlitelimab DPs (DP1 and DP2) | From Day1 up to Day92 (EOS)
  AUC after administration of a single SC dose of amlitelimab DP1 and DP 2

SECONDARY OUTCOMES:
Part 1 and Part 2: Incidence of adverse events (AE)/treatment-emergent adverse events (TEAEs) | From the signing of the informed consent form (ICF) up to Day92 EOS visit
  Incidence of AEs and TEAEs after administration of amlitelimab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Clinical Pharmacology of Miami-Site Number: 8400001, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM17597 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25329&tenant=MT_SNY_9011